CLINICAL TRIAL: NCT01165658
Title: Phase I Study of Hypofractionated Proton Radiation Therapy in Thoracic Malignancies
Brief Title: Study of Hypofractionated Proton Radiation Therapy in Thoracic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Requested by PI during yearly Continuing Review
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0164; NCI-2012-01780 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Non-small Cell Lung Cancer; Small Cell Lung Cancer; Carcinoid; Thymic Cancer; Lung Cancer
Keywords: non-small cell lung cancer; NSCLC; small cell lung cancer; SCLC; carcinoid; thymic cancer; lung cancer; radiation therapy; radiotherapy; proton therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoid Tumor; Thymus Neoplasms; Lung Neoplasms | interventions — Proton Therapy; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Therapy (Experimental): The radiation prescription dose ranges from 45 Gy in 3 Gy fractions to 60 Gy in 4 Gy fractions. Patients will be assigned to receive 1 of 3 doses of radiation therapy, based on when they joined the study. The first group of at least 3 participants will receive the lowest total radiation dose. If the first dose is tolerated well by the first group of participants in this study, then the next group of participants will receive the second, higher dose of radiation. If this dose is tolerated, then a third group will be treated at the highest dose.
  Interventions: Radiation: Proton Therapy

INTERVENTIONS:
Radiation: Proton Therapy — The regimen of 45 Gy in 15 fractions will be delivered as a baseline, and then the fraction size will be escalated in two different intervals of 0.5 Gy each, with the ultimate dose being 60 Gy in 4 Gy fractions.
  Other Names: Radiation; XRT; Radiotherapy

SUMMARY:
The goal of this clinical research study is to study the safety of giving larger daily doses of proton radiation therapy than the standard dose levels given to treat lung cancer. Researchers want to find the highest daily dose of proton radiation that can be given without having to stop therapy due to side effects.

DETAILED DESCRIPTION:
Proton Therapy:

Proton therapy is a type of radiation that is designed to lower the amount of radiation given to the healthy tissue around the tumor by using a more focused beam of radiation.

Radiation Dose Levels:

If you are found to be eligible to take part in this study, you will be assigned to receive 1 of 3 doses of radiation therapy, based on when you joined the study. The first group of at least 3 participants will receive the lowest total radiation dose. If the first dose is tolerated well by the first group of participants in this study, then the next group of participants will receive the second, higher dose of radiation. If this dose is tolerated, then a third group will be treated at the highest dose.

Practice Visit:

You will have a "practice" radiation visit to plan how the radiation will be given, about 1 week before therapy. This practice visit should take about 1-2 hours. At this visit, you will have a CT scan of the chest that will be used by the study staff to plan your proton therapy. A mold (made of the type of material used for casts) will also be made around your body that will be used to help you remain still during radiation therapy. Marks will be made on your skin to help position your body correctly for the radiation therapy. These marks may be permanent or temporary. If temporary marks are washed off, they will be replaced.

Proton Therapy Visits:

About 1 week after the practice radiation visit, you will begin receiving radiation therapy. At each visit, you will lie down in the mold of your body that was made at the practice visit, and you will be lined up for radiation therapy using the marks made on your skin at the practice visit.

You will receive radiation therapy every weekday (Monday-Friday) for about 3 weeks. Each radiation session should last about 45-60 minutes.

Study Tests:

Each week while you are receiving radiation therapy, you will be asked about any side effects you may be having. Your medical history will be recorded, and you will have a physical exam. If your doctor thinks it is needed, blood (about 2 tablespoons each time) will be drawn for routine tests, and/or you may have CT scans to check the status of the tumor.

Length of Therapy:

You will receive proton radiation therapy for about 3 weeks. The radiation therapy will be stopped early if the disease gets worse or intolerable side effects occur.

Follow-up Visits:

About 6 weeks after your last dose of proton radiation, you will have a CT scan of the chest (with a contrast agent, if possible) and a physical exam.

About 3 months after the first follow-up visit you will have a physical exam, lung function tests, and either a PET/CT scan or CT scan of the chest to check the status of the disease.

Long-term Follow-up:

Every 3 months for the first 2 years after you finish proton therapy, every 6 months for the next 3 years, and 1 time every year after that, you will be asked to return to the clinic for follow-up tests. These tests may include lung function tests, imaging scans (such as a CT or PET/CT scan), and/or an ECG. This will be up to your doctor.

This is an investigational study. At this time, it is considered investigational to give proton radiation therapy at the dose schedule used in this study. This schedule is being used for research purposes only.

Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented NSCLC, SCLC, thymic tumors, or carcinoid tumors
2. Patients not receiving concurrent chemotherapy
3. Patients that are eligible for concurrent treatment with biologic agents (epidermal growth factor receptor [EGFR] or vascular endothelial growth factor [VEGF] inhibitors) will be eligible for the study.

Exclusion Criteria:

1. Prior radiotherapy to the chest
2. Life expectancy <6 months
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07-16 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Hypofractionated Proton Therapy | 1 month after completion of radiation therapy
  Dose-limiting toxicity (DLT) defined as any CTCAE v4.0 grade 4 complication of esophagus or skin, or any grade 3 or higher complications of other organ systems (i.e. lung, liver, kidney, or GI tract), unless these complications are deemed to be related to those of esophagus. DLT assessed within 1 month of completion of radiation therapy. MTD defined as highest dose for which probability of toxicity is closest to 25%.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gomez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org